CLINICAL TRIAL: NCT06180070
Title: Randomized, Two-way, Two-period, Single Oral Dose, Open-label, Crossover, Bioequivalence Study to Compare Ibuprofen/ Paracetamol Tablets (200mg Ibuprofen/ 500mg Paracetamol) Versus Nuromol® Tablets (200mg Ibuprofen/ 500mg Paracetamol) in Healthy Subjects Under Fasting Condition
Brief Title: Bioequivalence Study to Compare Ibuprofen/ Paracetamol Tablets (200mg Ibuprofen/ 500mg Paracetamol) Versus Nuromol® Tablets (200mg Ibuprofen/ 500mg Paracetamol)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1246-2023
Record Dates: First submitted 2023-12-05; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Migraine; Headache; Backache
MeSH Terms: conditions — Migraine Disorders; Headache; Back Pain | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibuprofen/ Paracetamol tablets (Experimental): Ibuprofen/ Paracetamol tablets (200mg Ibuprofen/ 500mg Paracetamol)
  Interventions: Drug: Ibuprofen/ Paracetamol tablets; Drug: Nuromol® tablets
- Nuromol® tablets (Active Comparator): Nuromol® tablets (200mg Ibuprofen/ 500mg Paracetamol)
  Interventions: Drug: Ibuprofen/ Paracetamol tablets; Drug: Nuromol® tablets

INTERVENTIONS:
Drug: Ibuprofen/ Paracetamol tablets — 1 tablet of 200mg Ibuprofen/ 500mg Paracetamol
Drug: Nuromol® tablets — 1 tablet of 200mg Ibuprofen/ 500mg Paracetamol

SUMMARY:
Randomized, two-way, two-period, single oral dose, open-label, crossover, bioequivalence study to compare Ibuprofen/ Paracetamol tablets (200mg Ibuprofen/ 500mg Paracetamol) versus Nuromol® tablets (200mg Ibuprofen/ 500mg Paracetamol) in healthy subjects under fasting condition.

ELIGIBILITY:
Inclusion Criteria

* The subject is Caucasian & aged between eighteen to fifty years (18 - 50), both inclusive.
* The subject is within the limits for his height & weight as defined by the body mass index range (18.5 - 30.0 Kg/m2).
* The subject is willing to undergo the necessary pre- & post- medical examinations set by this study.
* The results of medical history, vital signs, physical examination & conducted medical laboratory tests are normal as determined by the clinical investigator.
* The subject tested negative for Hepatitis B (HBsAg), Hepatitis C (HCVAb) and human immunodeficiency virus (HIVAb).
* There is no evidence of psychiatric disorder, antagonistic personality, and poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* The subject is able to understand and willing to sign the informed consent form.
* The subject has normal cardiovascular system & normal ECG recording with normal QT interval corrected for heart rate according to Bazett's formula.
* The subject's kidney and liver (AST & ALT enzymes) function tests are within normal range. (Creatinine is accepted if below the reference range after being evaluated by the clinical investigator as clinically not significant).
* For female subjects: negative serum pregnancy test and the woman is using two reliable contraception methods and should be non-lactating.

Exclusion Criteria

* The subject is a heavy smoker (more than 10 cigarettes per day).
* The subject has suffered an acute illness one week before dosing.
* The subject has a history of or concurrent abuse of alcohol.
* The subject has a history of or concurrent abuse of illicit drugs.
* The subject has a history of hypersensitivity and/or contraindications to the study drug and any related compounds such as Aspirin or other NSAIDs.
* The subject has been hospitalized within three months before the study or during the study.
* The subject is on diet (for example subject is vegetarian.)
* The subject has consumed caffeine or xanthine containing beverages or foodstuffs within two days before dosing and until 23 hours after dosing in either study period.
* The subject has taken a prescription medication within two weeks or even an over the counter product (OTC) within one week before dosing in each study period and any time during the study, unless otherwise judged acceptable by the clinical investigator.
* The subject has taken grapefruit/ orange containing beverages or foodstuffs within seven (7) days before dosing and any time during the study.
* The subject has been participating in any clinical study (e.g. pharmacokinetics, bioavailability and bioequivalence studies) within the last 80 days prior to the present study.
* The subject has donated blood within 80 days before first dosing.
* The subject has a history or presence of cardiovascular, pulmonary, renal, hepatic, gastrointestinal, hematological, endocrinal, immunological, dermatological, neurological, musculoskeletal or psychiatric diseases.
* The subject has consumed drugs, foodstuffs or supplements that may affect pharmacological or pharmacokinetic properties of Ibuprofen/ Paracetamol (for example: NSAIDs, corticosteroids, methotrexate, sulfamethoxazole, ACE inhibitors, beta blockers, diuretics, chlorpropamide, Chlorpropamide, quinolone antibiotics, macrolide group antibiotics, Cholestyramine, heparin and warfarin) two weeks before dosing, during the study and two weeks after dosing.
* The subject has a history of, or active, peptic ulceration, esophagitis, gastritis, gastrointestinal bleeding or perforation, any gastrointestinal disorders or chronic inflammatory disease (e.g. ulcerative colitis, crohn's disease).
* The subject has any signs/symptoms of an infection such as fever or pain.
* The subject has a history of blood clotting disorders.
* Subjects having systemic lupus erythematous or other mixed connective tissue disease.
* Female subjects planning to become pregnant.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Maximum concentration obtained (Cmax) | 23 hours
  two-sided 90% CI for the test to reference ratio of the population means is within 80.00 - 125.00% for each of the Ln-transformed data Cmax
AUC from time 0 to last collection time t (AUC0-t) | 23 hours
  two-sided 90% CI for the test to reference ratio of the population means is within 80.00 - 125.00% for each of the Ln-transformed data AUC0-t

SECONDARY OUTCOMES:
AUC from time 0 to infinity (AUC0-∞) | 23 hours
  Descriptive Statistics
Time to reach maximum concentration Cmax (Tmax) | 23 hours
  Descriptive Statistics

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Gürpınar, Study Director — Humanis Saglık
Locations (1):
- ACDIMA Biocenter, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No